CLINICAL TRIAL: NCT04598295
Title: A Randomized, Double Blind, Placebo-controlled Study to Evaluate the Impact of a Multi-strain Synbiotic on Fecal Metagenomic Stability, Gut Barrier Integrity, and Metabolic Output of the Gut Microbiota
Brief Title: SH-DS01 on Fecal Metagenomic Stability
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Seed Health (Industry)
Responsible Party: Principal Investigator, Judy Nee, Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019P-000274
Record Dates: First submitted 2020-08-31; First posted 2020-10-22 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- microbial consortia (DS-01) (Experimental): DS-01 is a rationally defined microbial consortia consisting of 24 strains across 12 species, with polyphenolic and phenolic prebiotic bioactive compounds. Participants will be instructed to take 2 capsules daily for the duration of the trial.
  Interventions: Drug: DS-01
- placebo (Placebo Comparator): Placebo capsules for DS-01 will contain rice flour matched for color and texture in an identical outer capsule shell. Participants will be instructed to take 2 capsules daily for the duration of the trial.
  Interventions: Drug: DS-01

INTERVENTIONS:
Drug: DS-01 — synbiotic
  Other Names: SEED synbiotic

SUMMARY:
This is a randomized, double blind, Phase 1 study. There will be a 12-week comparison of the safety of DS-01 versus placebo with a secondary outcome measure of the efficacy in a cohort of 100 men or women with IBS with constipation. 50 IBS-C or IBS-M patients will receive DS-01 (Daily Synbiotic, once daily) for 12 weeks, while 50 IBS-C or IBS-M patients will receive the placebo (once daily). Safety is a paramount concern in the study design and will be monitored carefully throughout the study. Study subjects will also receive extensive education on use of the synbiotic.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is a chronic functional gastrointestinal disorder that generates a significant health care burden and is the most commonly diagnosed gastrointestinal condition. Nearly 12% of all patients in the United States seek medical care in primary care practice for IBS and it accounts for 3.1 million ambulatory care visits and 5.9 million prescriptions annually.

The pathophysiology of IBS is distinctly broad compared to other gastrointestinal conditions and includes abnormalities involving motility, visceral sensation, brain-gut interaction, and distress. Though patients with IBS often have a heterogeneous symptom profile, the predominant theme is the presence of abdominal pain or discomfort that is usually relieved by defecation. Host factors such as genetics, immune function, and psychological status, as well as environmental factors such as stress, recent infection, or treatment with antibiotics, could predispose to the development of chronic IBS symptoms. Due to a myriad of contributing factors, a single cause of IBS remains enigmatic. Despite the urgent need to develop better therapies, the high range of placebo response has made clinical trials challenging, ranging from 16.0 to 71.4% with a population-weighted average of 40.2%.

Recent studies have also shown alterations in gut immune response, and a disrupted intestinal and colonic microbiome in association with IBS. The current working hypothesis is that abnormal microbiota activate mucosal innate immune responses, which increase epithelial permeability, activate nociceptive sensory pathways, and dysregulate the enteric nervous system. Targeting the microbiota and gastrointestinal tract with live organisms is a promising approach, yet previous trials have yielded limited success due to empiric strain selection, small population size, and inadequate trial design to control for a high placebo response.

This protocol aims to assess the impact of a multi-strain consortia of 24 commensal organisms across 12 species with extensive strain-specific in vivo data, assessing a range of gastrointestinal symptoms without negatively altering the naive gut microbiota. High-throughput shotgun DNA sequencing will provide opportunity for '-omics'-based analyses of the gut microbiota, which can be augmented by the metabolite profiles resulting from total microbial activity in the gut. Since many of these metabolites are bioeffector molecules acting upon the host, such analysis can provide a direct measure of the consequences of microbial activity in the gut and provide a novel integrated data set for patients with IBS. Recruited subjects will also use a smart-phone application to report day to day gastrointestinal symptoms, a patient-centric hallmark of this chronic gut condition.

Probiotics are live microorganisms with a vast array of therapeutic potential for gastrointestinal disease. Several probiotics strains have shown beneficial outcomes in constipation-predominant IBS (IBS-C) patients, especially as an adjunct to conventional treatment. However, a number of controversial issues regarding the roles of probiotics in pathogenesis of IBS-C remain to be clarified, including precise mechanism of action.

This protocol aims to assess the impact of a mix of 24-beneficial strains on individual gastrointestinal symptoms specifically in a cohort of subjects with IBS-C or IBS-M.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be willing and able to give informed assent/ consent for participation in the study
* Patient must be willing and able (in the PI's opinion) to comply with all study requirements.
* Patient must be a premenopausal female or male aged 18 and older.
* Patient must have a documented history of IBS that is not completely controlled by current IBS drugs.
* Patient must have a score of ≥150 on the IBS-SSS at screening.
* Patient must have no clinically relevant (in the judgment of the PI) abnormal blood laboratory levels at screening or randomization.
* The clinician will assess eligibility as per the Rome IV criteria (Recurrent abdominal pain or discomfort at least 1 day/week in the last 3 months associated with two or more of the following: Improvement with defecation. Onset associated with a change in frequency of stool).

Exclusion Critieria:

* Patient has clinically significant unstable medical conditions other than IBS.
* Patient has had clinically relevant symptoms or a clinically significant illness in the four weeks prior to screening or randomization.
* Patient has clinically significant laboratory values (in the PI's opinion).
* Patient is currently using or has in the past used recreational or medicinal cannabis, or synthetic cannabinoid based medications (including Sativex®) or supplements (including hemp oil/extracts) within one month prior to study entry and is unwilling to abstain for the duration for the study.
* Patient has consumed any probiotic product three days prior to screening and/or is unwilling to abstain from consuming these during the study.
* Intake of antibiotics in the past 1-month (i.e. penicillin, amoxicillin, cephalexin (Keflex), erythromycin (E-Mycin), clarithromycin (Biaxin), azithromycin (Zithromax), ciprofloxacin (Cipro), levofloxacin (Levaquin), ofloxacin (Floxin), co-trimoxazole (Bactrim), trimethoprim (Proloprim), tetracycline (Sumycin or Panmycin), doxycycline (Vibramycin), gentamicin (Garamycin), or tobramycin (Tobrex). The supplement in the present study may have a minor interaction with these medications.
* Patient has any known or suspected hypersensitivity to pomegranate, pine, or mushrooms, or any of the excipients of the Supplement Synbiotic Product (SSP).
* Patients of child bearing potential unless willing to ensure that they use effective contraception, for example, oral contraception, double barrier, intra-uterine device, during the study and for three months thereafter.
* Patients who are pregnant, lactating, or planning pregnancy during the course of the study and for three months thereafter.
* Patients who have been part of a clinical trial involving any investigational product in the previous six months.
* Any other significant disease or disorder which, in the opinion of the PI, may either put the patient at risk because of participation in the study, may influence the result of the study, or affect the patient's ability to participate in the study.
* Patient has significantly impaired hepatic function at Visit 1 (Alanine aminotransferase (ALT) >5 × upper limit of normal (ULN) or bilirubin >2 × ULN) OR the ALT or Aspartate aminotransferase (AST) >3 × ULN and the bilirubin >2 × ULN (or international normalized ratio >1.5).
* Obesity (BMI > 30)
* Implantable device such as heart pacemaker.
* Patients unwilling to abstain from donation of blood during the study.
* History of inflammatory bowel disease.
* History of diverticulosis.
* History of cardiovascular disease.
* History of kidney/liver/serious infection.
* History of diabetes or other hormone diseases.
* History of abdominal surgery.
* Currently suffering from high blood pressure.
* Following a physical examination, the patient has any abnormalities that, in the opinion of the investigator would prevent the patient from safe participation in the study.
* There are plans for the patient to travel outside the USA during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of DS-01 treatment vs placebo | 12 weeks
  measure of reported adverse events

SECONDARY OUTCOMES:
Metagenomic Signature Change in Synbiotic group 1 | 12 weeks
  Participants displaying a change in metagenomic signatures resulting in increased representation from baseline of Bifidobacterium longum, or Prevotella intermedia or Bacteroides helcogenes or Akkermansia muciniphila or decreased representation of Blautia hansenii in subjects with IBS-C receiving DS-01 as greater than placebo treated subjects.
Metagenomic Signature Change in Synbiotic group 2 | 12 weeks
  Participants displaying a change in metagenomic signatures resulting in an increased representation from baseline of Alistipes finegoldii or Faecalibacterium prausnitzii or Akkermansia muciniphila or decreased representation from baseline of Blautia obeum in subjects with IBS-M receiving DS-01 greater than placebo treated subjects.
Improvement by ≥ 15% in one or more individual IBS symptoms: abdominal pain, bloating, bowel movement difficulty, or stool consistency. | 12 weeks
  Self-reported in a Symptom Tracker app to track disease progression in real-time
Abdominal pain responder | 12 weeks
  Percentage of responders in the intervention group who report a ≥ 20% reduction in average daily worst abdominal pain scores compared to placebo.
CSBM Responder | 12 weeks
  Percentage of responders in subjects with IBS-C receiving DS-01 who report an increase from baseline of 1 complete spontaneous bowel movement (CSBM) per week for at least 6 weeks compared to placebo
Global Improvement in IBS | 12 weeks
  Measured with one question with 7 possible answers: (1) much worse, (2) moderately worse, (3) slightly worse, (4) unchanged, (5) slightly better, (6) moderately better, or (7) much better.
Adequate Relief | 12 weeks
  A higher proportion of subjects in the DS-01 intervention group with Adequate Relief of Global IBS Symptoms for ≥ 30% in the intervention duration compared to the placebo group
VSI responder | 12 weeks
  A higher proportion of subjects with improvement ≥ 30% in Visceral Sensitivity Index score in the DS-01 intervention group compared to the placebo group.
Maintenance or increase of diversity within the DS-01 treatment group [baseline-Day 84] | 12 weeks
  Microbiota composition will be identified through fecal samples for total genomic DNA extraction in participants supplemented with DS-01 or placebo. Metagenomic sequencing will yield a total observable species count and maintenance will be defined as a change in total observed species less than or equal to 20% as compared to the total observed species count at baseline.

OTHER OUTCOMES:
Exploratory endpoint 1 | 12 weeks
  Increase in tryptamine, SCFA, and hypoxanthine production in IBS-C, changes in serine protease, LPS, or calprotectin in the DS-01 intervention group compared to the placebo group.
Exploratory endpoint 2 | 12 weeks
  Change in plasma intestinal fatty acid binding protein (I-FABP), zonulin, LPS-binding protein, soluble CD14, cytokines

CONTACTS AND LOCATIONS:
Overall Officials: Anthony J Lembo, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No